CLINICAL TRIAL: NCT00348868
Title: Miami Buprenorphine HIV Care Integration Project
Brief Title: Buprenorphine HIV Care Integration Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: HRSA/Maternal and Child Health Bureau (U.S. Federal Agency); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Margaret A. Fischl, M.D., Unversity of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A007
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Last update posted 2008-03-18 (Estimated); Status verified 2007-04

CONDITIONS: HIV Infection; Opioid-Related Disorders
Keywords: HIV Infection; Opioid dependence; DSM-IV criteria for opioid dependence
MeSH Terms: conditions — HIV Infections; Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): enhanced behavioral motivation counseling
  Interventions: Behavioral: enhanced behavioral motivation counseling; Behavioral: Motivational counseling
- 2 (Active Comparator)
  Interventions: Behavioral: Standard counseling

INTERVENTIONS:
Behavioral: enhanced behavioral motivation counseling
  Arms: 1
Behavioral: Motivational counseling
  Arms: 1
Behavioral: Standard counseling
  Arms: 2

SUMMARY:
A007 is a randomized, two-arm study evaluating the effectiveness of standard drug addiction counseling with buprenorphine/naloxone to enhanced motivational drug counseling with buprenorphine/naloxone for the treatment for opioid addiction in an integrated and nonintegrated HIV care setting.

DETAILED DESCRIPTION:
DESIGN: A007 is a randomized, two-arm study evaluating the effectiveness of standard drug addiction counseling with buprenorphine/naloxone to enhanced motivational drug counseling with buprenorphine/naloxone for the treatment for opioid addiction in an integrated and nonintegrated HIV care setting.

DURATION: Subjects will participate in this study for approximately 48 weeks. Chart abstractions will continue for up to four years.

SAMPLE SIZE: This study will enroll 60 subjects (30 per arm) over 72 weeks.

POPULATION: HIV-1 infected opioid dependent men and women ≥18 years of age who initiate buprenorphine for the treatment of opioid dependence and who are receiving primary care for HIV-1 infection.

STRATIFICATION: Subjects will be stratified at screening based on HIV care setting (integrated HIV care vs. nonintegrated HIV care)

INTERVENTON At entry subjects will be randomized to one of the following:

ARM A: Standard drug addiction counseling + buprenorphine / naloxone

ARM B: Enhanced behavioral motivation counseling + buprenorphine / naloxone

The three primary outcomes are:

1. Cessation of illicit opioid use
2. Reduction in high risk behavior
3. Improved HIV therapy adherence

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* Receiving or seeking outpatient HIV care
* Seeking outpatient treatment for opioid dependence and be willing to take buprenorphine
* Meets DSM-IV criteria for opioid dependence, and be willing to stop illicit opioid use and be experiencing early symptoms of opioid withdrawal at the time that buprenorphine is given
* Men and women age ≥ 18 years
* Women of reproductive potential must have a negative serum or urine pregnancy test result available within 7 days prior to initiating buprenorphine
* Within 30 days: (SGOT), ALT (SGPT), and alkaline phosphatase <=5 X ULN, Total bilirubin <= 2.5 x ULN

Exclusion Criteria:

* Serious medical problem
* Acute and/or severe psychiatric conditions
* High dose methadone (>30 mg/day)
* Documented co-dependence on alcohol and/or benzodiazepines, barbiturates
* Chronic pain management requiring opioids
* Pregnancy or breast-feeding
* Imprisonment or involuntary incarceration in a medical facility for psychiatric or physical

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The three primary outcomes are Cessation of illicit opioid use, Reduction in high risk behavior and Improved HIV therapy adherence | week 48

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Fischl, M.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami AIDS Clinical Reserach Unit, Miami, Florida, United States